CLINICAL TRIAL: NCT00550030
Title: Prospective, Randomized Half-side Study on the Efficacy of UVB-311nm Phototherapy in Patients With Psoriasis Undergoing Etanercept Treatment
Brief Title: Etanercept Plus UVB-311nm Phototherapy in Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Peter Wolf, MD, Professor of Bioimmunotherapy, Medical University of Graz
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-257 ex 05/06
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; UVB radiation; Biologics; Etanercept; PASI
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- left/right (Experimental): half-body comparison
  Interventions: Radiation: UVB-311nm radiation; Other: No treatment

INTERVENTIONS:
Radiation: UVB-311nm radiation — UVB-311nm radiation randomized to one body half given 3 times a week for 6 weeks; the other body half remains UV-non-irradiated.
  Other Names: Narrow band UVB radiation
Other: No treatment — no UV exposure

SUMMARY:
Etanercept, a biological antipsoriatic drug with anti-tumor-necrosis factor (TNF) activity has been approved for the treatment of moderate to severe psoriasis. However, in a substantial portion of cases etanercept does not induce reduction in psoriasis area and severity index (PASI) of 75% or greater, now being considered as gold standard for treatment efficacy. In this study the researchers aim to determine in a randomized half-side comparison, whether additional narrowband UVB-311nm phototherapy accelerates and improves the therapeutic efficacy of etanercept.

DETAILED DESCRIPTION:
Patients with moderate to severe psoriasis who have received a standard dose of etanercept (50 mg or 25 mg s.c. twice weekly) for at least 6 weeks without a PASI reduction of 75% or greater qualify for the study. Etanercept is continued and UVB-311nm phototherapy is added at 6 weeks or thereafter on a randomized body half (left or right; head exempt) 3 x per week until complete response (defined as reduction in PASI to < 3) for a maximum of another 6 weeks (until week 12). PASI score and patient disease score is assessed weekly; patient life quality score at week 0, 6, and 12; all scores at follow-up visits at month 3, 6, and 12. Paired statistical testing (T-test or Wilcoxon) for differences in PASI and patient disease and life quality scores is done; Fischer exact test is applied to determine differences in complete remission, PASI reduction > 90%, > 75%, and/or 50% between body sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe psoriasis who have received a standard dose of etanercept (50 mg or 25 mg s.c. twice weekly) for at least 6 weeks without a PASI reduction of 75% or greater

Exclusion Criteria:

* Pregnancy or lactation
* Presence of or history of malignant skin tumors
* Dysplastic melanocytic nevus syndrome
* Antinuclear antibodies (ds-DNA, Ro/SSA, La/SSB)
* Autoimmune disorders such as Lupus erythematosus or Dermatomyositis
* Photosensitive diseases such as porphyria, chronic actinic dermatitis, Xeroderma pigmentosum, basal cell nevus syndrome, and others
* General poor health status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Reduction of PASI (psoriasis activity score index) | prospective

SECONDARY OUTCOMES:
Patient disease and life quality score | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Dept. of Dermatology, Medical University of Graz, Graz, Austria
Locations (1):
- Medical University of Graz, Department of Dermatology, Graz, Austria